CLINICAL TRIAL: NCT04152980
Title: Pentoxifylline Dose Optimization in Preterm Neonatal Late Onset Sepsis
Brief Title: Pentoxifylline Dose Optimization in Neonatal Sepsis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Sinno H.P. Simons, Neonatologist, Erasmus Medical Center
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: OZBS32.18194
Record Dates: First submitted 2019-06-21; First posted 2019-11-06 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Neonatal Late Onset Sepsis
Keywords: Pentoxifylline; preterm infants; sepsis treatment; dose optimization
MeSH Terms: conditions — Neonatal Sepsis | interventions — Pentoxifylline

STUDY DESIGN:
Intervention Model Description: Prospective dose optimizing study using a step-up and step-down model. In order to find the optimal dose, the infusion of pentoxifylline in different dosages will be studied, next to antibiotics with 3 patients per dosage. The first 3 patients will receive a dose of 5 mg/k/h for 6 h per day, comparable to the dose that has been used before in trials. Upward or downward dose adjustments for the following cohort of 3 patients will be considered. If the dose is effective, the next 3 patients will receive a lower dose, in order to find the lowest effective dose. After the dose optimization study an additional cohort of 10 patients will be treated with the determined optimal dose as a validation of this dose.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Pentoxifylline therapy 2,5 mg/kg/h for 3 hours. (Experimental): This is a dose optimization study, different dosages will be tested, the lowest dosage that will be tested is 2,5 mg/kg/h for 3 hours every 24 hours for 3 to 6 days. The decision to prolong therapy after 3 days of therapy is made by the treating physician, depending on the clinical state of the patient and the severity of disease.
  Interventions: Drug: Pentoxifylline
- Pentoxifylline therapy 2,5 mg/kg/h for 6 hours (Experimental): The second lowest dosage that will be tested is 2,5 mg/kg/h for 6 hours every 24 hours for 3 to 6 days. The decision to prolong therapy after 3 days of therapy is made by the treating physician, depending on the clinical state of the patient and the severity of disease.
  Interventions: Drug: Pentoxifylline
- Pentoxifylline therapy 5 mg/kg/h for 6 hours. (Experimental): The third lowest dosage, is the start dosage and the dosage that is already used in other clinical studies: 5 mg/kg/h for 6 hours every 24 hours for 3 to 6 days. The decision to prolong therapy after 3 days of therapy is made by the treating physician, depending on the clinical state of the patient and the severity of disease.
  Interventions: Drug: Pentoxifylline
- Pentoxifylline therapy 5 mg/kg/h for 12 hours. (Experimental): The fourth dosage that is tested is 5 mg/kg/h for 12 hours every 24 hours for 3 to 6 days. The decision to prolong therapy after 3 days of therapy is made by the treating physician, depending on the clinical state of the patient and the severity of disease..
  Interventions: Drug: Pentoxifylline
- Pentoxifylline therapy 5 mg/kg/h for 18 hours. (Experimental): The fifth dosage that is tested is 5 mg/kg/h for 18 hours every 24 hours for 3 to 6 days. The decision to prolong therapy after 3 days of therapy is made by the treating physician, depending on the clinical state of the patient and the severity of disease.
  Interventions: Drug: Pentoxifylline
- Pentoxifylline therapy 5 mg/kg/h for 24 hours. (Experimental): The sixth dosage that is tested is 5 mg/kg/h for 24 hours every 24 hours for 3 to 6 days. The decision to prolong therapy after 3 days of therapy is made by the treating physician, depending on the clinical state of the patient and the severity of disease.
  Interventions: Drug: Pentoxifylline

INTERVENTIONS:
Drug: Pentoxifylline — The intervention consists of intravenously administered pentoxifylline. Pentoxifylline , a methylxanthine, is an off patent drug for neonates and currently registered for peripheral artery disease treatment in adults. Pentoxifylline acts as a cyclic adenosine monophosphate(cAMP)-phosphodiesterase inhibitor that suppresses tumor necrosis factor alfa (TNF-α) and modulates important parts of the inflammatory response and also reduces the production of other inflammatory cytokines, such as IL-1α, IL-6, and IL-8.
  Other Names: Trental

SUMMARY:
Sepsis is a very important cause of death and morbidity in preterm infants. There are strong indications that preterm neonates with sepsis could benefit, next to antibiotics, from treatment with pentoxifylline (PTX). Knowledge about optimal dosing is however limited. This study is a dose optimization study using a step-up and step-down model. In order to find the optimal dose, the infusion of pentoxifylline in different dosages will be studied, next to antibiotics with 3 patients per dosage. After the dose optimization study an additional cohort of 10 patients will be treated with the found dosage as a validation of the dose.

DETAILED DESCRIPTION:
Rationale: Sepsis is a very important cause of death in preterm infants. Survival from sepsis is often related to severe short and long term morbidity. Despite optimal antibiotic treatment, immaturity of the immune system in preterm neonates causes this severe sepsis related mortality and morbidity. There are strong indications that preterm neonates with sepsis could benefit, next to antibiotics, from treatment with pentoxifylline. Pentoxifylline which is registered for adults with intermittent claudication, is already used in preterm neonates with sepsis. Knowledge about optimal dosing is however limited.

Objective: The main objective is to determine in what optimal dose pentoxifylline should be used in preterm infants suffering from sepsis. Previous clinical studies have already indicated the safety of the drug in preterm infants.

Study design: Dose optimisation study in preterm born infants with late onset sepsis and increased inflammation. In this study different dosages will be evaluated, with dosage step-up and step-down in every 3 patients. Starting dose will be the dose as described in all previous studies. Around 30 included neonates are expected to be needed to determine the optimal dose using this study design. Subsequently, The optimal dose will be validated in 10 preterm neonates.

Study population: Preterm born neonates with a gestational age below 30 weeks and suspected late onset sepsis and relevant inflammation are eligible for inclusion. To quantify inflammation, an interleukin-6 above 500 pg/mL and/ or a C- reactive protein above 50 mg/L is needed at initiation of pentoxifylline therapy.

Intervention: The intervention consists of intravenously administered pentoxifylline.

Main study parameters/endpoints: Primary outcome is the optimal dose of pentoxifylline. Optimized pentoxifylline dosage needs to be related with adequate biochemical response, adequate clinical response and no severe side effects/adverse drug reaction. In each patient it is determined if the patient has an adequate pentoxifylline dosage. The dosage is considered to be adequate if the biochemical response is adequate and the clinical outcome is adequate with no severe side effects. When 3 patients are treated with a certain dosage, a decision will be made whether to increase or decrease the dosage for the next 3 patients. If the dosage was considered inadequate (at least 2 patients in whom the dosage was inadequate) the dosage for the next patients will be increased. If the dosage was considered adequate( (at least 2 patients in whom the dosage was adequate) the dosage for the next patients will be decreased. Secondary endpoints include further understanding the inflammatory and immunological changes of preterm infants during sepsis with pentoxifylline treatment by measuring metabolomic biomarkers of the signalling and peroxidised lipid platform and 91 inflammatory proteomics.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Pentoxifylline is already used at our neonatal intensive care unit for patients with sepsis, but data on the dose/response curve do not exist. Pentoxifylline has already been shown to have beneficial effects in humans and animal models of sepsis, especially in preterm infants. A meta-analysis showed that pentoxifylline increases the survival of preterm infants suffering from sepsis and suggests that pentoxifylline is well tolerated. No severe side effects have been detected in previous studies or in clinical practice of preterm infants. A therapeutic gain for participants of the study is expected because of the expected benefits from optimized pentoxifylline treatment. Improved outcome of neonatal sepsis is expected. During the study a limited amount of additional blood will be collected either from arterial lines or during routine blood drawing. No extra heelsticks or venipunctures will be performed for the study. A maximum amount of 3% of the total blood volume is used for research purposes in a 4 weeks period. No further additional burden is expected

ELIGIBILITY:
Inclusion Criteria:

* Preterm born neonates with gestational age <30 weeks
* Suspected of late onset sepsis with blood drawn for blood culture and inflammatory biomarkers
* IL-6 > 500 pg/mL and/or CRP > 50 mg/L

Exclusion Criteria:

* pentoxifylline therapy cannot be started within 24 hours of start of antibiotic treatment.
* Major congenital defect (e.g. congenital heart disease, pulmonary, or gastrointestinal anomalies).
* IL-6 values exceeding 25000 pg/mL at time of onset. High IL-6 values represent severe episodes of sepsis and high IL-6 values are associated with high mortality rates.
* Already participated in this trial during an earlier episode of late onset sepsis.
* PH below 7 in two consecutive blood samples, with at least 1 hour between the blood samples, at start of sepsis episode.

Max Age: 30 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2020-01-12 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Adequate pentoxifylline dose | 3 days
  Adequate pentoxifylline doses are determined by 3 co-primary outcome variables:
  * Adequate biochemical response: CRP will be measured in blood at time of onset and 24 , 48 and 72 hours after onset. An area under the curve (AUC) will be calculated for each patient. An area under the curve below the 25th percentile of an historical cohort is considered to be adequate.
  * Adequate clinical outcome: if a patient has one of the following criteria, clinical outcome is considered inadequate: mortality, necrotizing enterocolitis greater than Bell stage 3, pH below 7 in 2 consecutive blood samples with at least 1 hour between the 2 samples after start of sepsis treatment and/or the need to start NO therapy with indication pulmonary hypertension after start of sepsis treatment.
  * No severe side effects/adverse drug reaction

SECONDARY OUTCOMES:
The levels of 91 inflammatory Olink proteomics markers measured in blood plasma and sepsis | If possible at 3 days old, 1 hour after sepsis onset, 6, 24, 48 hours after onset and at 7 days after sepsis onset.
  The inflammatory panel from Olink Proteomics will be used (link: https://www.olink.com/products/inflammation/) to measure 91 inflammatory proteomics will be measured in blood plasma during sepsis treatment. Olink proteomics are measured in Normalized Protein eXpression (NPX) (link: https://www.olink.com/question/what-is-npx/).
  The authors want is to further understand the inflammatory and immunological changes of preterm infants during sepsis with pentoxifylline treatment. This analyses will be exploratory, seeing that proteomics haven't been frequently used in neonatal sepsis (research). The aim is to find differential proteomic patterns among patients with gram negative sepsis, gram positive sepsis, culture negative sepsis or no infection. The authors will report proteomic patterns associated with sepsis.
The levels of metabolomic biomarkers of the signalling and peroxidised lipid platform measured in blood plasma and sepsis | If possible at 3 days old, 1 hour after sepsis onset, 6, 24, 48 hours after onset and at 7 days after sepsis onset.
  Metabolomics of the signalling and peroxidised lipid platform will be measured in blood plasma. The authors want to further understand the inflammatory and immunological changes of preterm infants during sepsis with pentoxifylline treatment. This platform covers the following classes of metabolomics:
  * Eicosanoids / Oxylipins
  * Endocannabinoids
  * Isoprostanes
  * Nitro fatty acids
  * Lysophopholipids & Sphingosine-1-phosphate
  * Polyunsaturated free fatty acids
  * Bile acids
  The aim is to find differential metabolomics patterns among patients with gram negative sepsis, gram positive sepsis, culture negative sepsis or no infection. The authors will report metabolomic patterns associated with sepsis. Metabolomics measurements are performed using mass spectrometry.
Pentoxifylline and metabolites levels in blood plasma during sepsis treatment | 3 days after start of pentoxifylline treatment
  Pentoxifylline concentrations will be analyzed in a pharmacokinetic model and will be integrated with pharmacodynamics data(biochemical response, side effects) and covariates(post menstrual age, weight, morbidity, etc). The authors will report effective pentoxifylline and metabolites concentrations (µg/ml) and concentrations (µg/ml) that might result in side-effects.
The levels of 91 inflammatory Olink proteomics markers measured in blood plasma and clinical outcome | If possible at 3 days old, 1 hour after sepsis onset, 6, 24, 48 hours after onset and at 7 days after sepsis onset.
  This will be exploratory, seeing that proteomics haven't been frequently used in neonatal sepsis (research). The predictive value of differential proteomic levels and changes in levels in predicting the clinical outcome (e.g. predicting hypotension, respiratory deterioration, etc.) will be evaluated. The inflammatory panel form Olink Proteomics will be used (link: https://www.olink.com/products/inflammation/). The authors will report proteomic levels and patterns in Normalized Protein eXpression (NPX) (link: https://www.olink.com/question/what-is-npx/).
The levels of metabolomic biomarkers of the signalling and peroxidised lipid platform measured in blood plasma and clinical outcome | If possible at 3 days old, 1 hour after sepsis onset, 6, 24, 48 hours after onset and at 7 days after sepsis onset.
  This will be exploratory, seeing that metabolomics haven't been frequently used in neonatal sepsis (research). The predictive value of differential metabolomic patterns in predicting the clinical outcome (e.g. predicting hypotension, respiratory deterioration, etc.) will be evaluated. Metabolomics of the signalling and peroxidised lipid platform will be measured in blood plasma. This platform covers the following classes of metabolomics:
  * Eicosanoids / Oxylipins
  * Endocannabinoids
  * Isoprostanes
  * Nitro fatty acids
  * Lysophopholipids & Sphingosine-1-phosphate
  * Polyunsaturated free fatty acids
  * Bile acids The authors will report metabolomics levels and patterns by measuring metabolomics using mass spectrometry.
The levels of 91 inflammatory Olink proteomics markers measured in blood plasma and pentoxifylline and metabolites levels in blood plasma during sepsis treatment | If possible at onset of sepsis and 24 and 48 hours after onset of sepsis
  Associations between the proteomic levels and pentoxifylline exposure will be explored by visual inspection (i.e. scatter plots) and statistical comparisons as needed. Pentoxifylline exposure will be reported by pentoxifylline and metabolites concentrations (µg/ml) and proteomic levels will be reported in Normalized Protein eXpression (NPX) (link: https://www.olink.com/question/what-is-npx/).
The levels of metabolomic biomarkers of the signalling and peroxidised lipid platform measured in blood plasma and pentoxifylline and metabolites levels in blood plasma during sepsis treatment | If possible at onset of sepsis and 24 and 48 hours after onset of sepsis
  Associations between the metabolomic biomarkers of the signalling and peroxidised lipid platform and pentoxifylline exposure will be explored by visual inspection (i.e. scatter plots) and statistical comparisons as needed. This platform covers the following classes of metabolomics:
  * Eicosanoids / Oxylipins
  * Endocannabinoids
  * Isoprostanes
  * Nitro fatty acids
  * Lysophopholipids & Sphingosine-1-phosphate
  * Polyunsaturated free fatty acids
  * Bile acids
  Pentoxifylline exposure will be reported by pentoxifylline and metabolites concentrations (µg/ml) and metabolomics levels by measuring metabolomics using mass spectrometry.

CONTACTS AND LOCATIONS:
Overall Officials: Sinno Simons, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (2):
- Erasmus MC Sophia Children's Hospital, Rotterdam, Netherlands
- University Hospital Poznan, Poznan, Poland

IPD SHARING:
Plan to Share IPD: Yes
The investigators have made a Data management plan in DMPonline in collaboration with local datamanager Dr. A Ham.
  The investigators plan to publish in an open access journal There is a management plan considering making data findable, accessible and intraoperable and reusable.
Supporting Information: Study Protocol, CSR, Analytic Code
Time Frame: Protocol, Statistical Analysis Plan and Informed Consent Form will be shared after the protocol has been approved by the medical ethical committee.
Access Criteria: The data management plan is shared in a public area. The investigators intend to share our data after our clinical study report is published. Sharing of data will only occur after permission is given by the investigators.
URL: https://dmponline.dcc.ac.uk/public_plans

REFERENCES:
- [Background] Neuner P, Klosner G, Schauer E, Pourmojib M, Macheiner W, Grunwald C, Knobler R, Schwarz A, Luger TA, Schwarz T. Pentoxifylline in vivo down-regulates the release of IL-1 beta, IL-6, IL-8 and tumour necrosis factor-alpha by human peripheral blood mononuclear cells. Immunology. 1994 Oct;83(2):262-7. PMID 7835945
- [Background] Mandell GL. Cytokines, phagocytes, and pentoxifylline. J Cardiovasc Pharmacol. 1995;25 Suppl 2:S20-2. doi: 10.1097/00005344-199500252-00005. PMID 8699856
- [Background] Windmeier C, Gressner AM. Pharmacological aspects of pentoxifylline with emphasis on its inhibitory actions on hepatic fibrogenesis. Gen Pharmacol. 1997 Aug;29(2):181-96. doi: 10.1016/s0306-3623(96)00314-x. PMID 9251897
- [Background] Schroer RH. Antithrombotic potential of pentoxifylline. A hemorheologically active drug. Angiology. 1985 Jun;36(6):387-98. doi: 10.1177/000331978503600608. PMID 3927788
- [Background] Yang S, Zhou M, Koo DJ, Chaudry IH, Wang P. Pentoxifylline prevents the transition from the hyperdynamic to hypodynamic response during sepsis. Am J Physiol. 1999 Sep;277(3):H1036-44. doi: 10.1152/ajpheart.1999.277.3.H1036. PMID 10484426
- [Background] Zeni F, Pain P, Vindimian M, Gay JP, Gery P, Bertrand M, Page Y, Page D, Vermesch R, Bertrand JC. Effects of pentoxifylline on circulating cytokine concentrations and hemodynamics in patients with septic shock: results from a double-blind, randomized, placebo-controlled study. Crit Care Med. 1996 Feb;24(2):207-14. doi: 10.1097/00003246-199602000-00005. PMID 8605790
- [Background] Pammi M, Haque KN. Pentoxifylline for treatment of sepsis and necrotizing enterocolitis in neonates. Cochrane Database Syst Rev. 2015 Mar 9;(3):CD004205. doi: 10.1002/14651858.CD004205.pub3. PMID 25751631
- [Background] Haque KN, Pammi M. Pentoxifylline for treatment of sepsis and necrotizing enterocolitis in neonates. Cochrane Database Syst Rev. 2011 Oct 5;(10):CD004205. doi: 10.1002/14651858.CD004205.pub2. PMID 21975745
- [Derived] Kurul S, Taal HR, Flint RB, Mazela J, Reiss IKM, Allegaert K, Simons SHP. Protocol: Pentoxifylline optimal dose finding trial in preterm neonates with suspected late onset sepsis (PTX-trial). BMC Pediatr. 2021 Nov 18;21(1):517. doi: 10.1186/s12887-021-02975-8. PMID 34794420
- See also: Olink Proteomics Inflammation Panel — https://www.olink.com/products/inflammation/
- See also: Olink Proteomics NPX unit of measurement — https://www.olink.com/question/what-is-npx/